CLINICAL TRIAL: NCT03512522
Title: A Pain Self-management Program for Older Adults: Online vs. Workbook Delivery
Brief Title: Pain Self-management Program for Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Regina (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2018-004
Record Dates: First submitted 2018-04-18; First posted 2018-04-30 (Actual); Last update posted 2019-11-20 (Actual); Status verified 2019-11

CONDITIONS: Chronic Pain; Depression; Anxiety
Keywords: chronic pain; pain self-management; remote delivery; workbook; online
MeSH Terms: conditions — Chronic Pain; Depression; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: A patient preference randomized controlled trial (RCT) will be used for this study. Participants will be randomly assigned to be enrolled in the online group or workbook group, or be placed on a twelve-week wait list control, which will serve as a control group to control for the influence of time on symptom change between groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Online Group (Experimental): An 8-week remotely-delivered pain self-management program tailored to older adults that have been experiencing pain for at least three months. Participants randomized to the Online Group will receive access to the course on the computer (online). A researcher will act as a guide who provides general support and encouragement, as opposed to a clinician who would offer comprehensive therapy. The guide will aim to contact participants weekly via telephone for approximately 5 to 10 minutes.
  Interventions: Behavioral: Online Group
- Workbook Group (Experimental): An 8-week remotely-delivered pain self-management program tailored to older adults that have been experiencing pain for at least three months. Participants randomized to the Workbook Group will receive access to the course in a printed (workbook) format. A researcher will act as a guide who provides general support and encouragement, as opposed to a clinician who would offer comprehensive therapy. The guide will aim to contact participants weekly via telephone for approximately 5 to 10 minutes.
  Interventions: Behavioral: Workbook Group
- Wait List Control Group (No Intervention): Participants who are randomly allocated to the wait list control group will be provided access to the course after the twelve-week period has passed.

INTERVENTIONS:
Behavioral: Online Group — An 8-week remotely-delivered pain self-management program tailored to older adults that will be delivered in an online format.
  Arms: Online Group
Behavioral: Workbook Group — An 8-week remotely-delivered pain self-management program tailored to older adults that will be delivered in a printed (workbook) format.
  Arms: Workbook Group

SUMMARY:
It is well documented that severe pain is more common in older adults than it is younger persons. Of concern, older adults may not have access to traditional face-to-face self-management programs, which are recognized to be valuable in chronic pain management. Access to effective self-management approaches is particularly important for older adults who may have mobility limitations or live in remote areas, or have difficulty accessing health care services. The development of effective pain self-management programs for older adults who cannot access traditional psychological interventions is of significant importance. Internet self-management programs have the potential to address pain undermanagement. As technology advances, the digital divide between the older and younger demographic continues to progress. Given the known difficulties with treatment access, the purpose of this study is to explore the efficacy and acceptability of a remotely-delivered chronic pain self-management program tailored to older adults, the Pain Course, when delivered in online and workbook formats. The program was previously shown to be effective among younger persons but has not been tested with older adults.

DETAILED DESCRIPTION:
The program is delivered through a secure platform administered by the Online Therapy Unit for Service Education and Research at the University of Regina. Using a patient preference randomized control trial (RCT) design, participants (n = 120) will be enrolled in either the online group or workbook group, or to a wait list control group. The content of both programs will be identical and contain 5 core lessons, which participants will be encouraged to work through over an 8-week period. By exploring the efficacy of an online vs. workbook group, the results from this study may serve as a stepping-stone for improved self-management of chronic pain in older adults.

A patient preference randomized controlled trial (RCT) was chosen for this study. The goal is to have most participants accept randomization by emphasizing they are equally acceptable, so only those with a very strong preference or no access to Internet aren't randomized. According to the preliminary power analysis, a total of 120 participants will be randomly assigned to be enrolled in the online group or workbook group, or be placed on a twelve-week wait list control, which will serve as a control group to control for the influence of time on symptom change between groups.

ELIGIBILITY:
Inclusion Criteria:

* are residents of Canada
* are 65 years of age or older
* report experiencing pain for more than three months
* are not experiencing very severe symptoms of depression or anxiety
* have regular access to a computer and the internet
* are proficient in writing and speaking the English language

Exclusion Criteria:

* high suicide risk
* concerns about online therapy
* not present in the country during treatment
* are younger than 65 years of age

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 121 (Actual)
Dates: Start 2018-02-23 (Actual); Primary Completion 2019-04-20 (Actual); Study Completion 2019-04-20 (Actual)

PRIMARY OUTCOMES:
Change in the impact of pain in several areas of life | baseline, 8 weeks, 3 months
  Measured by Pain Disability Index (PDI)
Change in depression | baseline, 8 weeks, 3 months
  Measured by Geriatric Depression Scale-30 (GDS-30)
Change in anxiety | baseline, 8 weeks, 3 months
  Measured by Generalized Anxiety Disorder Scale 7-Item (GAD-7)
Change in chronic pain severity | baseline, 8 weeks, 3 months
  Measured by Brief Pain Inventory (BPI)

SECONDARY OUTCOMES:
Change in beliefs about one's ability to perform every day tasks regardless of chronic pain | baseline, 8 weeks, 3 months
  Measured by Pain Self-Efficacy Questionnaire (PSEQ)
Change in fear of movement or re-injury | baseline, 8 weeks, 3 months
  Measured by TAMPA Scale of Kinesiophobia (TSK)
Change in acceptance of chronic pain | baseline, 8 weeks, 3 months
  Measured by Chronic Pain Acceptance Questionnaire (CPAQ-8)
Change in tendency to amplify the threat value of constant pain | baseline, 8 weeks, 3 months
  Measured by Pain Catastrophizing Scale (PCS)
Treatment satisfaction | 8 weeks
  Measured by Treatment Satisfaction Questions (TSQ) used in Pain Course

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Hadjistavropoulos, Principal Investigator — University of Regina; Heather Hadjistavropoulos, Principal Investigator — University of Regina
Locations (1):
- University of Regina, Regina, Saskatchewan, Canada

IPD SHARING:
Plan to Share IPD: No